CLINICAL TRIAL: NCT04002115
Title: Clofarabine Pre-conditioning Followed by Hematopoietic Stem Cell Transplant With Post-Transplant Cyclophosphamide for Non-remission Acute Myeloid Leukemia
Brief Title: Clofarabine Pre-conditioning Followed by Stem Cell Transplant for Non-remission AML
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated due to low accrual
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Seema Naik, MD, Associate Professor of the Penn State Cancer Institute, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-011
Record Dates: First submitted 2019-06-24; First posted 2019-06-28 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Clofarabine; Haploidentical stem cell transplantation; matched and mismatched unrelated donors; Non-remission AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine; fludarabine; fludarabine phosphate; Busulfan; Whole-Body Irradiation; Cyclophosphamide; Granulocyte Colony-Stimulating Factor; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: Dose de-escalation: Enrollment will begin at 30 mg/m2 to analyze any grade 4-5 organ toxicities as defined in Section 12.2. If the trial is stopped due to excessive toxicities, then dose de-escalation to 20 mg/m2 will occur for the next cohort of participants. For each participant, the observation period is from start of treatment through post-transplant day +30. Adverse effects will be continuously monitored as patients are enrolled. The trial will be stopped when the toxicity rate exceeds 20% with a posterior probability of 80% and a margin of no more than 5%. This leads to the following stopping rule: the trial will be stopped if 2 of the first 3 subjects experience grade 4-5 organ toxicity, or 3 out of 6, 4 out 9, 5 out of 12, 6 out of 16, or 7 out 19.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Clofarabine 30 mg/m^2 (Experimental): Day -14 through Day -10 Clofarabine 30 mg/m^2, Day - 9 Day of rest, Day - 8 Day of rest, Day - 7 Day of rest, Day - 6 Fludarabine 40 mg/m^2 IV and Busulfan 3.2 mg/kg IV (Regimen A, Fludarabine 24 mg/m^2 IV and Cyclophosphamide 14.5 mg/kg IV for Regimen B), Day - 5 Fludarabine 40 mg/m^2 IV and Busulfan 3.2 mg/kg IV (Regimen A, Fludarabine 24 mg/m^2 IV and Cyclophosphamide 14.5 mg/kg IV for Regimen B), Day - 4 Fludarabine 40 mg/m^2 IV(Regimen A, Fludarabine 24 mg/m^2 IV for Regimen B), Day - 3 Fludarabine 40 mg/m^2 IV(Regimen A, Fludarabine 24 mg/m^2 IV for Regimen B), Day - 2 Day of Rest, Day -1 Total Body Irradiation 200 cGys, Day 0 stem cell transplant infusion, Day +1 Day of rest, Day +2 Day of rest, Day +3 Cyclophosphamide 50 mg/kg IV, Day +4 Cyclophosphamide 50 mg/kg IV, Day +5 Start G-CSF, Tacrolimus, and MMF.
  Interventions: Drug: Clofarabine; Drug: Fludarabine; Drug: Busulfan; Procedure: Total Body Irradiation (TBI); Drug: Cyclophosphamide; Drug: Granulocyte Colony-Stimulating Factor; Drug: Tacrolimus; Drug: Cellcept

INTERVENTIONS:
Drug: Clofarabine — Clofarabine to be administered pre-stem cell transplant infusion ("Day 0") once a day for 5 days total.
  Other Names: Clolar
Drug: Fludarabine — Fludarabine will be administered once a day for 4 days as part of the transplant conditioning regimen.
  Other Names: Fludara
Drug: Busulfan — Busulfan will be administered once a day for 2 days as part of the transplant conditioning regimen.
  Other Names: Busulfex
Procedure: Total Body Irradiation (TBI) — TBI will be administered at a dose of 200cGys on Day -1 prior to transplant
  Other Names: TBI
Drug: Cyclophosphamide — Cyclophosphamide will be given once a day for 2 days after the transplant infusion.
  Other Names: Cytoxan
Drug: Granulocyte Colony-Stimulating Factor — G-CSF will be administered to subjects starting on Day +5 and will continue as clinically indicated
  Other Names: Filgrastim G-CSF
Drug: Tacrolimus — Tacrolimus will be administered to subjects starting on Day +5 and will continue as clinically indicated
  Other Names: Prograf
Drug: Cellcept — Mycophenolate Mofetil will be administered to subjects starting on Day +5 and will continue as clinically indicated
  Other Names: Mycophenolate Mofetil (MMF)

SUMMARY:
The Investigators would like to study the incidence of complete remission (CR) at day +30 after Clofarabine followed by haploidentical transplant. The conditioning regimen used is Fludarabine, Busulfan (2 doses) or cyclophosphamide (2 doses) and Total Body Irradiation (TBI) with post transplant cyclophosphamide for patients with Acute Myeloid Leukemia (AML) who are not in remission prior to considering allogeneic transplant with haploidentical donors.

DETAILED DESCRIPTION:
Approximately 30-40% of patients with acute myeloid leukemia (AML) experience induction failures. In these patients who do not achieve remission with two cycles of standard induction therapies, the probability of achieving remission with subsequent inductions is limited. Hematopoietic stem cell transplantation (HSCT) is the only curative option for these patients, but high relapse rate and transplant-related mortality often preclude them to proceed to transplant. Thus, AML not in remission at time of HSCT remains a huge unmet need in current HSCT practice, particularly if the patient does not have a Human Leukocyte Antigen (HLA)-matched donor identified by the time of two induction failures.

Salvage chemotherapy with clofarabine appears to be another promising option in relapsed and refractory AML. Clofarabine is a second-generation purine nucleoside analog with substantial single-agent activity in adult patients with AML. It is an effective immunosuppressive agent and several trials have shown the feasibility of conditioning with clofarabine-based regimen.

In the past, a conditioning regimen of clofarabine with busulfan (4 doses) has been successfully used prior to allogeneic stem cell transplantation for non-remission AML with day +30 complete remission rates were 90-100%. However, these patients were transplanted with HLA matched donors. This study will examine those patients undergoing transplantation from haploidentical related donor or matched and mismatched unrelated donors.

Achieving a long-term remission is clearly the goal of AML treatment. The investigators would like to propose a protocol for non-remission AML and expand the patient population to older than 55 years of age as well as those who relapsed after initial allogeneic transplant to improve enrolling patients in the near future. The investigators have many patients achieving remission but for those without remission, clofarabine preconditioning may be a reliable protocol to bring these patients into the early complete remission.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic criteria of AML, induction failure without having achieved remission after at least 2 attempts at induction chemotherapy, or relapsed after any complete remission (CR).
2. 18 to 75 years of age.
3. Planned or scheduled to receive an allogeneic HSCT from haploidentical related donors, matched and mismatched unrelated donors.
4. All organ function testing should be done within 28 days of study registration.

   * Performance status: Karnofsky ≥ 70% (Appendix A).
   * Cardiac: LVEF ≥ 50% by MUGA or echocardiogram.
   * Pulmonary: FEV1 and FVC ≥ 50% predicted, DLCO (corrected for hemoglobin) ≥ 50% of predicted.
   * Renal: Creatinine clearance (CrCl) ≥ 60 mL/min/1.73 m2
   * Hepatic: Serum bilirubin ≤1.5 x upper limit of normal (ULN); (AST)/(ALT) ≤ 2.5 x ULN; Alkaline phosphatase ≤ 2.5 x ULN.
5. Both men and women need to use an approved method of birth control and/or abstinence due to unknown risks to the fetus.

Exclusion Criteria:

1. Acute promyelocytic leukemia (APL)
2. Known history of non-compliance with medication regimens, scheduled clinic visits, or self-care.
3. In the opinion of the investigator, no appropriate caregivers identified.
4. HIV1 (Human Immunodeficiency Virus-1) or HIV2 positive
5. Active Hepatitis B and Hepatitis C orepatitis positive serology including HBsAg, hepatitis B core antibody, and hepatitis C antibody. Hepatitis B surface antibody positive due to vaccination or natural immunity are permitted.
6. In the opinion of the physician investigator, uncontrolled medical or psychiatric disorders.
7. Uncontrolled infections requiring treatment within 14 days of registration.
8. Active central nervous system (CNS) leukemia.
9. Cord blood transplant excluded.
10. Prior allogeneic HSCT within last 6 months.
11. Patients with >= grade 2 acute GVHD.
12. Patients with >=moderate chronic GVHD.
13. Pregnant or Breastfeeding. Women of child bearing potential (WCBP) are required to have a negative serum or urine pregnancy test prior to initiation of conditioning regimen.
14. Haploidentical related donors who are positive for DSA ≥ 5000 MFI by solid phase microarray method (Luminex).
15. Any patient with steroid dose more than 10 mg/day within a week of registration .
16. Autoimmune disorder requiring any active immunosuppression therapy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema Naik, MD, Principal Investigator — Penn State Cancer Institute
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
At this time there is no plan to share IPD with other researchers outside of Penn State University

REFERENCES:
- See also: Penn State Cancer Institute — https://cancer.psu.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Both subjects were between age 56 and 75 years old, therefore they were assigned treatment of Regimen B.
Groups:
- Clofarabine 30 mg/m^2: Day -14 through Day -10 Clofarabine 30 mg/m^2, Day - 9 Day of rest, Day - 8 Day of rest, Day - 7 Day of rest, Day - 6 Fludarabine 24 mg/m^2 IV and Cyclophosphamide 14.5 mg/kg IV for Regimen B, Day - 5 Fludarabine 24 mg/m^2 IV and Cyclophosphamide 14.5 mg/kg IV, Day - 4 Fludarabine 24 mg/m^2 IV, Day - 3 Fludarabine 24 mg/m^2 IV, Day - 2 Fludarabine 24 mg/m^2 IV, Day -1 Total Body Irradiation 200 cGys, Day 0 stem cell transplant infusion, Day +1 Day of rest, Day +2 Day of rest, Day +3 Cyclophosphamide 50 mg/kg IV, Day +4 Cyclophosphamide 50 mg/kg IV, Day +5 Start G-CSF, Tacrolimus, and MMF.
  Clofarabine: Clofarabine to be administered pre-stem cell transplant infusion ("Day 0") once a day for 5 days total.
  Fludarabine: Fludarabine will be administered once a day for 5 days as part of the transplant conditioning regimen.
  Total Body Irradiation (TBI): TBI will be administered at a dose of 200cGys on Day -1 prior to transplant
  Cyclophosphamide: Cyclophosphamide will be given once a day for 2 days after the transplant infusion.
  Granulocyte Colony-Stimulating Factor: G-CSF will be administered to subjects starting on Day +5 and will continue as clinically indicated
  Tacrolimus: Tacrolimus will be administered to subjects starting on Day +5 and will continue as clinically indicated
  Cellcept: Mycophenolate Mofetil will be administered to subjects starting on Day +5 and will continue as clinically indicated
Period: Overall Study
Arm/Group | Clofarabine 30 mg/m^2
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Clofarabine 30 mg/m^2: Day -14 through Day -10 Clofarabine 30 mg/m^2, Day - 9 Day of rest, Day - 8 Day of rest, Day - 7 Day of rest, Day - 6, Fludarabine 24 mg/m^2 IV and Cyclophosphamide 14.5 mg/kg IV for Regimen B, Day - 5 Fludarabine 24 mg/m^2 IV and Cyclophosphamide 14.5 mg/kg IV for Regimen B, Day - 4 Fludarabine 24 mg/m^2 IV for Regimen B, Day - 3 Fludarabine 24 mg/m^2 IV for Regimen B, Day - 2 Fludarabine 24 mg/m^2 IV for Regimen B, Day -1 Total Body Irradiation 200 cGys, Day 0 stem cell transplant infusion, Day +1 Day of rest, Day +2 Day of rest, Day +3 Cyclophosphamide 50 mg/kg IV, Day +4 Cyclophosphamide 50 mg/kg IV, Day +5 Start G-CSF, Tacrolimus, and MMF.
Arm/Group | Clofarabine 30 mg/m^2
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR) Rate at Day 30 Post HSCT
Description: The CR rate at 30 days (Day +30) post stem cell transplant infusion
Time Frame: 30 days
Population: The CR rate at 30 days (Day +30) post stem cell transplant infusion was 2/2.
Measure: Number; unit: percentage of Participants
Groups:
- Clofarabine 30 mg/m^2: Day -14 through Day -10 Clofarabine 30 mg/m^2, Day - 9 Day of rest, Day - 8 Day of rest, Day - 7 Day of rest, Day - 6 Fludarabine 24 mg/m^2 IV and Cyclophosphamide 14.5 mg/kg IV for Regimen B, Day - 5 Fludarabine 24 mg/m^2 IV and Cyclophosphamide 14.5 mg/kg IV for Regimen B, Day - 4 Fludarabine 24 mg/m^2 IV for Regimen B, Day - 3 Fludarabine 24 mg/m^2 IV for Regimen B, Day - 2 Fludarabine 24 mg/m^2 IV for Regimen B, Day -1 Total Body Irradiation 200 cGys, Day 0 stem cell transplant infusion, Day +1 Day of rest, Day +2 Day of rest, Day +3 Cyclophosphamide 50 mg/kg IV, Day +4 Cyclophosphamide 50 mg/kg IV, Day +5 Start G-CSF, Tacrolimus, and MMF.
Arm/Group | Clofarabine 30 mg/m^2
Number analyzed (Participants) | 2
percentage of Participants | 100

2. Secondary Outcome: Non-relapse Related Mortality
Description: Determine the rate of non-relapse related mortality at 100 days post transplant (Day +100)
Time Frame: 100 days
Population: The rate of non-relapse related mortality at 100 days post transplant (Day +100) is 0/2.
Measure: Number; unit: percentage of Participants
Arm/Group | Clofarabine 30 mg/m^2
Number analyzed (Participants) | 2
percentage of Participants | 0

3. Secondary Outcome: Neutrophil Engraftment
Description: Rates of engraftment, defined as the first day of Absolute Neutrophil Count (ANC) greater than 500 for the first of three consecutive days
Time Frame: 1 year
Population: Rate of engraftment was 0/2.
Measure: Number; unit: percentage of Participants
Arm/Group | Clofarabine 30 mg/m^2
Number analyzed (Participants) | 2
percentage of Participants | 0

4. Secondary Outcome: Rate of Acute Graft-versus-host Disease (GVHD)
Description: The rate of any grade (1-4) of acute GvHD as measured from day of transplantation to Day +100 using the Glucksberg criteria.
Time Frame: 100 days
Population: The rate of any grade (1-4) of acute GvHD as measured from day of transplantation to Day +100 was 0/2.
Measure: Number; unit: percentage of Participants
Arm/Group | Clofarabine 30 mg/m^2
Number analyzed (Participants) | 2
percentage of Participants | 0

5. Secondary Outcome: Severity of Acute Graft-versus-host Disease (GVHD)
Description: The highest grade (1-4) of acute GvHD experienced by participants as measured from day of transplantation to Day +100 using the Glucksberg criteria
Time Frame: 100 days
Population: The highest grade (1-4) of acute GvHD experienced by participants as measured from day of transplantation to Day +100 was 0/2.
Measure: Number; unit: percentage of Participants
Arm/Group | Clofarabine 30 mg/m^2
Number analyzed (Participants) | 2
percentage of Participants | 0

6. Secondary Outcome: Rate of Chronic GVHD
Description: The rate of any grade (1-4) of Chronic GvHD as measured from Day +100 to Year 1 post-transplantation using the Glucksberg criteria.
Time Frame: 1 year
Population: The incidence of any grade (1-4) of Chronic GvHD as measured from Day +100 to Year 1 post-transplantation was 0/2.
Measure: Number; unit: percentage of Participants
Arm/Group | Clofarabine 30 mg/m^2
Number analyzed (Participants) | 2
percentage of Participants | 0

7. Secondary Outcome: Severity of Chronic GVHD
Description: The highest overall grade (1-4) of chronic GvHD experienced by participants as measured from Day +100 to Year 1 post-transplantation using the Glucksberg criteria
Time Frame: 1 year
Population: The highest overall grade (1-4) of chronic GvHD experienced by participants as measured from Day +100 to Year 1 post-transplantation was 0/2.
Measure: Number; unit: percentage of Participants
Arm/Group | Clofarabine 30 mg/m^2
Number analyzed (Participants) | 2
percentage of Participants | 0

ADVERSE EVENTS:
Time Frame: 1st subject: 10 months 2nd subject: 5 months
Groups:
- Clofarabine 30 mg/m^2: Day -14 through Day -10 Clofarabine 30 mg/m^2, Day - 9 Day of rest, Day - 8 Day of rest, Day - 7 Day of rest, Day - 6 Fludarabine 24 mg/m^2 IV and Cyclophosphamide 14.5 mg/kg IV for Regimen B, Day - 5, Fludarabine 24 mg/m^2 IV and Cyclophosphamide 14.5 mg/kg IV for Regimen B, Day - 4 Fludarabine 24 mg/m^2 IV for Regimen B, Day - 3 Fludarabine 24 mg/m^2 IV for Regimen B, Day - 2 Fludarabine 24 mg/m^2 IV for Regimen, Day -1 Total Body Irradiation 200 cGys, Day 0 stem cell transplant infusion, Day +1 Day of rest, Day +2 Day of rest, Day +3 Cyclophosphamide 50 mg/kg IV, Day +4 Cyclophosphamide 50 mg/kg IV, Day +5 Start G-CSF, Tacrolimus, and MMF.
Arm/Group | Clofarabine 30 mg/m^2
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine 30 mg/m^2 (N=2)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Multiorgan failure (General disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine 30 mg/m^2 (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (5)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Blood bilirubin increased (Investigations) | 2 (3)
Creatinine increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (5)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (4)
Nausea (Gastrointestinal disorders) | 2 (4)
Edema limbs (General disorders) | 1 (9)
Fatigue (General disorders) | 1 (2)
Fever (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Headche (Nervous system disorders) | 1 (5)
Lethargy (Nervous system disorders) | 1 (3)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2)
Weight gain (Investigations) | 2 (17)
Alkaline phosphatase increased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (3)
Hypophosphatemia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (2)
Tremor (Nervous system disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (5)
Hypotension (Vascular disorders) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1)
Increased bicarbonate level (Investigations) | 1 (2)
Abnormal EKG (Investigations) | 1 (1)
Increased BUN (Investigations) | 1 (5)
Increased RDW (Investigations) | 1 (1)
Increased specific gravity (Investigations) | 1 (1)
Hypoproteinemia (Investigations) | 1 (1)
Bladder wall thickening on CT abdomen (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to slow accrual, the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT04002115/Prot_SAP_000.pdf